CLINICAL TRIAL: NCT04429490
Title: Organochlorine Concentration in Adipose Tissue and Pancreatic Adenocarcinoma : a Case Control Study.
Brief Title: Organochlorine Concentration in Adipose Tissue and Pancreatic Adenocarcinoma
Acronym: PESTIPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PA20035
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2024-10

CONDITIONS: Carcinoma; Pancreatic Ductal
Keywords: Plant production products; risk factor; adipose tissue; organochlorine; pesticides
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group "Cases" (Experimental): patients with pancreatic adenocarcinoma
  Interventions: Other: Adipose tissue sampling during surgery and urine sampling
- Group "Controls" (Other): patients without pancreatic adenocarcinoma
  Interventions: Other: Adipose tissue sampling during surgery and urine sampling

INTERVENTIONS:
Other: Adipose tissue sampling during surgery and urine sampling — Adipose tissue sampling during surgery and urine sampling

SUMMARY:
Pancreatic adenocarcinoma represents more than 90% of pancreatic neoplasms. Around 14000 new cases of pancreatic adenocarcinoma are being diagnosed each year in France and about 8.6% in Grand Est region. National incidence has doubled for men and tripled for women between 1982 and 2012. Pancreatic adenocarcinoma is the deadliest digestive cancer, with only 7 to 8% all stages 5-year survival. It will become the second deadliest in Europe, behind bronchopulmonary cancer.

Several risk factors have been identified such as diabetes, tobacco, chronic pancreatitis or obesity. However, a mismatch exists between incidence forecasts and actual risk factors knowledge. Several hypothesis plead for an environnemental cause.

Plant protection products oncogenetic effects are known and have been proved to be responsible for tumors, including haematological malignancies. Its role in pancreatic carcinogenesis is still poorly studied and show heterogeneous results. They do not allow to conclude for causality. Organochlorines is a specific subset of plant protection product that store in lipids during lifetime.

The aim is to study association between organochlorine concentration in adipose tissue with pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Unicentric prospective case control study comparing organochlorine levels including patients diagnosed with a pancreatic adenocarcinoma undergoing a surgery allowing to collect an adipose tissue sample (10g).

Controls are adults with no pancreatic cancer (excluded by a 6 months old computed tomography excluding the probability of a pancreatic neoplasm), paired with cases upon age and body mass index, with a scheduled surgical procedure allowing to collect an adipose tissue sample without extending procedure length.

ELIGIBILITY:
inclusion criteria :

Cases :

* patients diagnosed with a pancreatic adenocarcinoma, all stages allowed
* undergoing a surgery allowing to take a 10 grams adipose tissue sample

Controls :

* patients without a pancreatic neoplasm on a 6 months old CT scan before inclusion
* undergoing a surgery allowing to take a 10 grams adipose tissue sample

exclusion criteria :

Cases :

* patients diagnosed with a pancreatic adenocarcinoma developed on IPMN or cystadenoma
* patient with a known genetic predisposition increasing pancreatic adenocarcinoma risk
* histopathology proof of a mixed neuroendocrine neoplasm
* no surgery allowing to take a 10 grams adipose tissue sample

Controls :

* patients with a pancreatic neoplasm on a 6 months old CT scan before inclusion
* no surgery allowing to take a 10 grams adipose tissue sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Adipose tissue organochlorine concentration | Day 0
  QuEChERS method to extract organochlorines Use of Agilent 7010 Detection limit : 10ng/g of adipose tissue

SECONDARY OUTCOMES:
Urine organochlorine concentration | Day 0
  Use of Agilent 7010 Detection limit : 0.1microg/L

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Result] Brugel M, Callon S, Carlier C, Amroun KL, Botsen D, Kianmanesh R, Perrier M, Piardi T, Renard Y, Rhaiem R, El Balkhi S, Bouche O. Association between pancreatic adenocarcinoma risk and concentration of organochlorine pesticides in adipose tissue and urine: A targeted-screening analysis case-control study (PESTIPAC). United European Gastroenterol J. 2024 Sep;12(7):951-959. doi: 10.1002/ueg2.12602. Epub 2024 Aug 8. PMID 39118264